CLINICAL TRIAL: NCT01088061
Title: Adipocytokines in Lean and Obese Women With and Without PCOS
Brief Title: Adipose Expression of Leptin, Adiponectin and IL-6 and Plasma Levels of Adipocytokines in Women With and Without Polycystic Ovary Syndrome (PCOS)
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Aarhus University Hospital (Other); Statens Serum Institut (Other)
Responsible Party: Copenhagen University Hospital, Hvidovre, Hospital
Other Study IDs: pcos0509
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2008-01

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fat biopsies, plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- lean women with PCOS
- Obese women with PCOS
- lean control women
- Obese control women

SUMMARY:
The purpose of the study was to investigate adipose expression and plasma levels of different adipocytokine, which may play a role in the pathophysiology of PCOS. The investigators investigated lean and obese women with and without PCOS.

ELIGIBILITY:
Inclusion Criteria:

* women with PCOS according to the Rotterdam criteria

Exclusion Criteria:

* other known diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Lean and obese women with and without PCOS, age 18-40 years.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2004-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Adipose expression of adipocytokines | From February 2004 -April 2006

SECONDARY OUTCOMES:
Plasma levels of adipocytokines | From February 2004-April 2006

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Fog Svendsen, MD, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark, Denmark